CLINICAL TRIAL: NCT03990051
Title: Treatment Safety and Efficacy Using Pro-ocular™ 1% for Chronic Ocular Graft-versus-host Disease (GvHD) Following Allogeneic Hematopoietic Stem Cell Transplantation.
Brief Title: Treatment Safety and Efficacy of Pro-ocular™ 1% for Chronic Ocular Graft Following Allogeneic HSCT.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glia, LLC (Industry)
Collaborators: ORA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: oGvHD-1
Record Dates: First submitted 2019-06-11; First posted 2019-06-18 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2024-11

CONDITIONS: Chronic Ocular Graft-versus-host Disease

STUDY DESIGN:
Intervention Model Description: The double-masked phase involves placebo controlled administration of study drug for 70 days or 10 weeks. Subsequently the placebo group will receive the active study drug of 42 days or 6 weeks. Long term open label phase to 27 months.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomized double-masked parallel treatment assignment will be made using a block design at the ratio of 2:1, study drug:placebo, (22 subjects:11 subjects). This 70-day double-masked phase will be followed by 6 weeks open-label active drug treatment of the subjects previously on placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pro-ocular™ (Experimental): Pro-ocular™ 1% topical gel applied dermally to forehead twice daily, morning and before bedtime.
  Interventions: Drug: Pro-ocular™ topical gel
- Placebo (Placebo Comparator): Vehicle topical gel without active ingredient applied dermally to forehead twice daily, morning and before bedtime.
  Interventions: Drug: Placebo topical gel

INTERVENTIONS:
Drug: Pro-ocular™ topical gel — Topical gel for forehead dermal application
  Arms: Pro-ocular™
Drug: Placebo topical gel — Topical gel for forehead dermal application
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of Pro-ocular™ 1% topical gel administered twice daily for 70 days in reducing or eliminating symptoms and signs of chronic ocular GvHD.

DETAILED DESCRIPTION:
Ocular graft versus host disease presents a most severe form of ocular surface disease that compromises quality of life of afflicted allogeneic hematopoietic transplantation patients.

A controlled study is necessary to verify findings obtained to date in isolated patients. Currently available ophthalmic solutions and suspensions, drugs and devices largely have not been effective in alleviating the suffering of chronic ocular GvHD patients. Thus, this is an unmet need that Pro-ocular™ topical gel can fulfill.

Potential benefits: Decrease or cessation of adverse ocular symptoms and signs of chronic ocular GvHD, reduction or elimination of the need for other topical ocular therapeutic treatments for chronic ocular GvHD, and restoration of quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female of any race, at least 18 years of age at Visit 1 Screening.
2. Has the diagnosis of chronic ocular GvHD.
3. Has an NIH Consensus Eye Score of at least 2.
4. On the GLIA Ocular Surface Disease Symptoms Questionnaire at Screening, has ocular discomfort at a severity score of moderate or more, and at least one other symptom at a severity of moderate or more.
5. One or more signs from the list of chronic ocular GvHD signs below
6. Has provided verbal and written informed consent.
7. Be able and willing to follow oral and written instructions, including participation in all study assessments and visits.

Exclusion Criteria:

1. Wearing scleral or contact lenses within the last month, or those who plan to start wearing scleral or contact lenses during the study.
2. Anticipate major changes in systemic GvHD management during study period.
3. Comorbidity with other severe or chronic eye conditions that in the judgment of the investigator will interfere with study assessments, such as but not limited to retinal detachment, recent ocular surgery, Bell's palsy, active trigeminal neuritis or trigeminal neuralgia.
4. Anticipate change of vision correction or anticipate any ocular procedures during study period.
5. A woman who is pregnant, nursing an infant, or planning a pregnancy.
6. A woman of childbearing potential who has a positive urine pregnancy test at Visit 1, or who does not use an adequate method of birth control throughout the study period.
7. Has a known adverse reaction and/or sensitivity to the study drug or its components.
8. Unwilling to cease the use of sunscreen on the forehead or eye area.
9. Intraocular pressure >22 mm Hg at screening visit with or without ongoing glaucoma treatment.
10. Currently enrolled in an investigational drug or device study for chronic ocular GvHD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghui K Luo, MD, PhD, Principal Investigator — Massachusetts Eye and Ear, Longwood
Locations (1):
- Massachusetts Eye and Ear Longwood, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Data may be shared with other investigators.

REFERENCES:
- [Result] Luo ZK, Domenech-Estarellas EA, Han A, Lee D, Khatri R, Wahl JL, Cutler C, Armand P, Antin JH, Koreth J, Gooptu M, Alyea EP, Soiffer RJ, Ho VT. Efficacy and Safety of 1% Progesterone Gel to the Forehead for Ocular Chronic Graft-versus-Host Disease. Transplant Cell Ther. 2021 May;27(5):433.e1-433.e8. doi: 10.1016/j.jtct.2021.02.008. Epub 2021 Feb 14. PMID 33942724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Double masked phase 10 weeks. Both Pro-ocular and Placebo groups received active treatment after 10 weeks for remainder of 2 years total from first dose..
Groups:
- Pro-ocular™: Pro-ocular™ 1% topical gel applied dermally to forehead twice daily, morning and before bedtime.
  Pro-ocular™ group received active for 2 years beginning with first dose. The first 10 weeks were masks, whereas the remaining time was open-label active.
- Placebo: Topical gel without active ingredient applied dermally to forehead twice daily, morning and before bedtime.
  Placebo group was dosed with placebo topical gel for the first 10 weeks, followed by open-label active for the remainder of 2 years from first dosing.
Period: Masked Period
Arm/Group | Pro-ocular™ | Placebo
Started | 22 | 11
Completed | 21 | 11
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: Long Term Period
Arm/Group | Pro-ocular™ | Placebo
Started | 21 | 11
Completed | 13 | 8
Not Completed | 8 | 3
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 7 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pro-ocular™: Pro-ocular™ 1% topical gel
- Placebo: Placebo topical gel
- Total: Total of all reporting groups
Arm/Group | Pro-ocular™ | Placebo | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (12.48) | 58.9 (13.20) | 60.9 (12.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 12
  Male | 13 | 8 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 22 | 11 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 21 | 9 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 22 | 11 | 33
Ocular Graft versus Host Diagnosis [Count of Participants; unit: Participants] | 22 | 11 | 33
Time of HSCT to oGvHD Diagnosis [Mean (Standard Deviation); unit: months] | 27.5 (22.5) | 40.0 (49.9) | 31.6 (33.8)
NIH Eye Score [Count of Participants; unit: Participants] — The NIH Eye Score is a scoring system used to measure the severity of dry eyes in patients with chronic ocular graft-versus-host disease (GVHD). The score ranges from 0-3, with 0 indicating no dry eye, 1 indicating mild dry eye, 2 indicating moderate dry eye, and 3 indicating severe dry eye.
  Participants
    Score 0-1 | 0 | 0 | 0
    Score 2 | 13 | 5 | 18
    Score 3 | 9 | 6 | 15
Concomitant artificial tears and gel [Count of Participants; unit: Participants] — Concomitant artificial tears and gel use
  Participants | 21 | 9 | 30
Concomitant ocular corticosteroid [Count of Participants; unit: Participants] — Concomitant ocular corticosteroid use.
  Participants | 15 | 8 | 23
Concomitant ocular ciclosporin [Count of Participants; unit: Participants] — Concomitant ciclosporin eye drops use.
  Participants | 2 | 2 | 4
Punctal plugs history [Count of Participants; unit: Participants] — Ever had punctal plugs inserted
  Participants | 18 | 11 | 29
Concomitant systemic anti-inflammatory [Count of Participants; unit: Participants] — Concomitant use of systemic anti-inflammatory medications
  Participants | 11 | 9 | 20

OUTCOME MEASURES:

1. Primary Outcome: Modified SANDE Questionnaire - Frequency, Change From Baseline
Description: Change in score from Baseline for worse eye. Score is 0-100 on a visual analog scale, higher values represent worse outcomes.
  Symptom Assessment iN Dry Eye Questionnaire. How often do eyes feel dry and/or irritated?
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Pro-ocular™: Pro-ocular™ 1% topical gel forehead BID
- Placebo: Placebo topical gel forehead tBID
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -22.00 (4.246) | -4.59 (6.009)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline, Active - Placebo; p = 0.0197, Mixed Models Analysis

2. Primary Outcome: Corneal Fluorescein Stain - Central, Change From Baseline
Description: Change in score from Baseline for worse eye. Fluorescein staining score in central corneal region recorded on visual analog scale 0-10, higher values represent worse outcomes.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Placebo topical gel forehead BID
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -0.90 (0.213) | 0.20 (0.304)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0039, Mixed Models Analysis

3. Secondary Outcome: Modified SANDE Questionnaire - Frequency, Change From Baseline
Description: as for outcome 1
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -31.75 (4.313) | -1.95 (6.009)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p < 0.0001, Mixed Models Analysis

4. Secondary Outcome: Modified SANDE Questionnaire - Frequency, Change From Baseline
Description: as for outcome 1
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -30.72 (4.313) | -2.18 (6.009)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0002, ANCOVA

5. Secondary Outcome: Corneal Fluorescein Stain - Central, Change From Baseline
Description: as for outcome 2
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Pro-ocular™: Pro-ocular™ 1% topical gel applied dermally to forehead twice daily
- Placebo: Placebo topical gel applied dermally to forehead twice daily
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -0.93 (0.216) | -0.01 (0.304)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0138, Mixed Models Analysis

6. Secondary Outcome: Corneal Fluorescein Stain - Central, Change From Baseline
Description: as for outcome 2
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.18 (0.216) | 0.06 (0.307)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0014, Mixed Models Analysis

7. Secondary Outcome: Modified SANDE Questionnaire - Global, Change From Baseline
Description: Change in score from Baseline for worse eye. Score is 0-100 on a visual analog scale, higher values represent worse outcomes.
  Symptom Assessment iN Dry Eye Questionnaire. How often do eyes feel dry and/or irritated? Global score is sqrt of Frequency x Severity.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -16.02 (4.063) | -3.78 (5.753)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0849, Mixed Models Analysis

8. Secondary Outcome: Modified SANDE Questionnaire - Global, Change From Baseline
Description: as for outcome 7
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -26.35 (4.128) | -5.64 (5.753)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0041, Mixed Models Analysis

9. Secondary Outcome: Modified SANDE Questionnaire - Global, Change From Baseline
Description: as for outcome 7
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -25.87 (4.128) | -1.04 (0.006)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0006, Mixed Models Analysis

10. Secondary Outcome: Corneal Fluorescein Stain - Total, Change From Baseline
Description: Change in score from Baseline for worse eye. Fluorescein staining score in Total comprise Central, Inferior and Superior regions, sum score 0-30, higher values represent worse outcomes.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -2.53 (0.527) | -0.23 (0.753)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0143, Mixed Models Analysis

11. Secondary Outcome: Corneal Fluorescein Stain - Total, Change From Baseline
Description: as for outcome 10
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -3.28 (0.537) | -1.35 (0.753)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0398, Mixed Models Analysis

12. Secondary Outcome: Corneal Fluorescein Stain - Total, Change From Baseline
Description: as for outcome 10
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -3.97 (0.537) | -1.54 (0.763)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = -3.97, Mixed Models Analysis

13. Secondary Outcome: Blurred Vision, Change From Baseline
Description: Change in score from Baseline for worse eye. Score measured from visual analog scale 0-10, higher values represent worse outcomes.
  Blurred vision symptom is reported by participant.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -2.07 (0.400) | 0.40 (0.568)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0005, Mixed Models Analysis

14. Secondary Outcome: Blurred Vision, Change From Baseline
Description: as for outcome 13
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -2.09 (0.404) | 0.39 (0.568)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0005, Mixed Models Analysis

15. Secondary Outcome: Blurred Vision, Change From Baseline
Description: as for outcome 13
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -2.23 (0.404) | -0.31 (0.568)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0067, Mixed Models Analysis

16. Secondary Outcome: Photophobia, Change From Baseline
Description: Change in score from Baseline for worse eye. Score is recorded on a visual analog scale 0-10, higher values represent worse outcomes.
  Sensitivity to light symptom is reported by participant.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.23 (0.432) | 0.18 (0.695)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0636, Mixed Models Analysis

17. Secondary Outcome: Photophobia, Change From Baseline
Description: as for outcome 16
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.68 (0.437) | 0.62 (0.613)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0028, Mixed Models Analysis

18. Secondary Outcome: Photophobia, Change From Baseline
Description: as for outcome 16
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.82 (0.437) | 0.01 (0.612)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0067, Mixed Models Analysis

19. Secondary Outcome: Lid Edema, Change From Baseline
Description: Change in score from Baseline for worse eye. Score on a visual analog scale 0-10, higher values represent worse outcomes.
  Lid edema is viewed by slit lamp without stain.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.73 (0.206) | -0.80 (0.293)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0105, Mixed Models Analysis

20. Secondary Outcome: Lid Edema, Change From Baseline
Description: as for outcome 19
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -2.21 (0.210) | -0.98 (0.293)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0010, Mixed Models Analysis

21. Secondary Outcome: Lid Edema, Change From Baseline
Description: as for outcome 19
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.72 (0.210) | -0.83 (0.293)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0155, Mixed Models Analysis

22. Secondary Outcome: Lid Erythema, Change From Baseline
Description: Change in score from Baseline for worse eye. Score on a visual analog scale 0-10, higher values represent worse outcomes.
  Lid erythema is viewed by slit lamp without stain.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.08 (0.224) | -0.13 (0.317)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0160, Mixed Models Analysis

23. Secondary Outcome: Lid Erythema, Change From Baseline
Description: as for outcome 22
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.53 (0.229) | -0.58 (0.317)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0117, Mixed Models Analysis

24. Secondary Outcome: Lid Erythema, Change From Baseline
Description: as for outcome 22
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.42 (0.229) | -1.27 (0.354)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.4649, Mixed Models Analysis

25. Secondary Outcome: Lid Margin Ulceration, Change From Baseline
Description: Change in score from Baseline for worse eye. Score on a visual analog scale 0-10, higher values represent worse outcomes.
  Lid margin ulceration is viewed by slit lamp without stain.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.14 (0.240) | -0.01 (0.341)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0082, Mixed Models Analysis

26. Secondary Outcome: Lid Margin Ulceration, Change From Baseline
Description: as for outcome 25
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.57 (0.245) | -0.59 (0.341)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0225, Mixed Models Analysis

27. Secondary Outcome: Lid Margin Ulceration, Change From Baseline
Description: as for outcome 25
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.85 (0.245) | -1.27 (0.354)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.1822, Mixed Models Analysis

28. Secondary Outcome: Conjunctival Hyperemia, Change From Baseline
Description: Change in score from Baseline for worse eye. Score on a visual analog scale 0-10, higher values represent worse outcomes.
  Conjunctival hyperemia is viewed by slit lamp without stain.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.50 (0.235) | -0.70 (0.333)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0515, Mixed Models Analysis

29. Secondary Outcome: Conjunctival Hyperemia, Change From Baseline
Description: as for outcome 28
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.75 (0.240) | -0.92 (0.333)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.044, Mixed Models Analysis

30. Secondary Outcome: Conjunctival Hyperemia, Change From Baseline
Description: as for outcome 28
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.72 (0.240) | -0.99 (0.333)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes of score from baseline; p = 0.083, Mixed Models Analysis

31. Secondary Outcome: Dryness, Change From Baseline
Description: Change in score from Baseline for worse eye. Score on a visual analog scale 0-10, higher values represent worse outcomes.
  Dryness symptom is reported by participant.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -2.48 (0.391) | -2.23 (0.554)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.7147, Mixed Models Analysis

32. Secondary Outcome: Dryness, Change From Baseline
Description: as for outcome 31
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -2.91 (0.398) | -2.76 (0.554)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.8251, Mixed Models Analysis

33. Secondary Outcome: Dryness, Change From Baseline
Description: as for outcome 31
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -3.67 (0.398) | -2.28 (0.554)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0435, Mixed Models Analysis

34. Secondary Outcome: Ocular Pain, Change From Baseline
Description: Change in score from Baseline for worse eye. Score on a visual analog scale 0-10, higher values represent worse outcomes.
  Ocular pain symptom is reported by participant.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.64 (0.310) | -0.29 (0.439)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0130, Mixed Models Analysis

35. Secondary Outcome: Ocular Pain, Change From Baseline
Description: as for outcome 34
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.53 (0.316) | -0.99 (0.439)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.3205, Mixed Models Analysis

36. Secondary Outcome: Ocular Pain, Change From Baseline
Description: as for outcome 34
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.86 (0.316) | -1.06 (0.499)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.1401, Mixed Models Analysis

37. Secondary Outcome: Airflow Sensitivity, Change From Baseline
Description: Change in score from Baseline for worse eye. Score on a visual analog scale 0-10, higher values represent worse outcomes.
  Airflow sensitivity symptom is reported by participant.
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.93 (0.401) | -0.68 (0.567)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison in changes in score from baseline; p = 0.0098, ANCOVA

38. Secondary Outcome: Airflow Sensitivity, Change From Baseline
Description: as for outcome 37
Time Frame: 6 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.69 (0.407) | -0.53 (0.583)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.1032, Mixed Models Analysis

39. Secondary Outcome: Airflow Sensitivity, Change From Baseline
Description: as for outcome 37
Time Frame: 10 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Pro-ocular™ | Placebo
Number analyzed (Participants) | 22 | 11
score on a scale | -1.76 (0.407) | -0.31 (0.567)
Statistical Analysis 1: Comparison: Pro-ocular™ vs Placebo; Test type: Superiority — Comparison of changes in score from baseline; p = 0.0389, Mixed Models Analysis

40. Other Pre Specified Outcome: Modified SANDE Questionnaire - Frequency
Description: Score on a visual analog scale 0-100, higher values represent worse outcomes. Symptom Assessment iN Dry Eye Questionnaire. How often do eyes feel dry and/or irritated?
Time Frame: 1 year
Population: The total number of participants were combined in one group for the 1 year analysis as all participants were dosed with active Pro-ocular after 10 weeks.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- Pro-ocular + Placebo Baseline: All participants combined as one group at baseline
- Pro-ocular + Placebo at 1 Year: All participants combined at 1 year as all were on active after 10 weeks
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
units on a scale | 82.03 (11.719) | 33.04 (27.517)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Score in 1 year compared to baseline; Test type: Other; p < 0.00001, t-test, 2 sided

41. Other Pre Specified Outcome: Modified SANDE Questionnaire - Frequency
Description: as for outcome 40
Time Frame: 2 years
Population: The total number of participants were combined in one group for the 2 year analysis as all participants were dosed with active Pro-ocular after 10 weeks.
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Groups:
- Pro-ocular + Placebo at 2 Years: All participants combined at 2 years as all were on active after 10 weeks
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
units on a scale | 82.03 (11.719) | 35.29 (27.637)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

42. Other Pre Specified Outcome: Modified SANDE Questionnaire - Global
Description: Score on a visual analog scale 0-100, higher values represent worse outcomes. Symptom Assessment iN Dry Eye Questionnaire. Global score is square root of how often do eyes feel dry and/or irritated x how severe are your symptoms of dryness and/or irritation?
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
units on a scale | 74.39 (16.620) | 32.63 (24.407)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Other; p < 0.00001, t-test, 2 sided

43. Other Pre Specified Outcome: Modified SANDE Questionnaire - Global
Description: as for outcome 42
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
units on a scale | 74.39 (16.620) | 31.04 (22.037)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

44. Other Pre Specified Outcome: Corneal Fluorescein Stain - Central
Description: Fluorescein staining score in central corneal region recorded on visual analog scale 0-10, higher values represent worse outcomes.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
units on a scale | 3.57 (2.779) | 1.12 (1.522)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Other; p = 0.0002, t-test, 2 sided

45. Other Pre Specified Outcome: Corneal Fluorescein Stain - Central
Description: as for outcome 44
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
units on a scale | 3.57 (2.779) | 0.77 (1.224)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p = 0.0001, t-test, 2 sided

46. Other Pre Specified Outcome: Corneal Fluorescein Stain - Total
Description: Fluorescein staining score Total for worse eye. Total comprise Central, Inferior and Superior regions, sum score 0-30, higher values represent worse outcomes.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
units on a scale | 11.52 (7.137) | 3.65 (3.289)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Other; p < 0.00001, t-test, 2 sided

47. Other Pre Specified Outcome: Corneal Fluorescein Stain - Total
Description: Fluorescein staining score Total for worse eye. Total comprises Central, Inferior and Superior regions, sum score 0-30, higher values represent worse outcomes.
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
units on a scale | 11.52 (7.137) | 2.81 (3.699)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

48. Other Pre Specified Outcome: Blurred Vision
Description: Score for worse eye, recorded on a visual analog scale 0-10, higher values represent worse outcomes.
  Blurred vision symptom is reported by participant.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
units on a scale | 7.59 (2.610) | 2.20 (2.582)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Superiority; p < 0.00001, t-test, 2 sided

49. Other Pre Specified Outcome: Blurred Vision
Description: as for outcome 48
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
units on a scale | 7.59 (2.610) | 1.66 (2.768)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

50. Other Pre Specified Outcome: Lid Edema
Description: Score for worse eye on a visual analog scale 0-10, higher values represent worse outcomes.
  Lid edema is scored by ophthalmologist using slit lamp biomicroscopy without staining.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
score on a scale | 3.74 (2.785) | 0.72 (0.995)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Other; p < 0.00001, t-test, 2 sided

51. Other Pre Specified Outcome: Lid Edema
Description: as for outcome 50
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
score on a scale | 3.74 (2.785) | 0.71 (1.085)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

52. Other Pre Specified Outcome: Lid Erythema
Description: Score for worse eye on a visual analog scale 0-10, higher values represent worse outcomes.
  Lid erythema is scored by ophthalmologist using slit lamp biomicroscopy without staining.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Groups:
- Pro-ocular + Placebo at 1 Year: All participants combined at 1 year all were on active after 10 weeks
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
score on a scale | 3.92 (2.738) | 1.17 (1.457)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Other; p = 0.0001, t-test, 2 sided

53. Other Pre Specified Outcome: Lid Erythema
Description: as for outcome 52
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Groups:
- Pro-ocular + Placebo at 2 Years: All participants combined at 2 years all were on active after 10 weeks
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
score on a scale | 3.92 (2.738) | 0.80 (1.144)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

54. Other Pre Specified Outcome: Lid Ulceration
Description: Score for worse eye on a visual analog scale 0-10, higher values represent worse outcomes.
  Lid ulceration is scored by ophthalmologist using slit lamp biomicroscopy without staining.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
score on a scale | 4.07 (2.289) | 1.14 (1.143)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Other; p < 0.00001, t-test, 2 sided

55. Other Pre Specified Outcome: Lid Ulceration
Description: as for outcome 52
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
score on a scale | 4.07 (2.289) | 0.42 (0.628)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

56. Other Pre Specified Outcome: Conjunctival Hyperemia
Description: Score for worse eye on a visual analog scale 0-10, higher values represent worse outcomes.
  Conjunctival hyperemia is scored by ophthalmologist using slit lamp biomicroscopy without staining.
Time Frame: 1 year
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 1 Year
Number analyzed (Participants) | 33 | 25
score on a scale | 3.67 (2.354) | 0.80 (1.238)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 1 Year; Test type: Other; p < 0.00001, t-test, 2 sided

57. Other Pre Specified Outcome: Conjunctival Hyperemia
Description: as for outcome 56
Time Frame: 2 years
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pro-ocular + Placebo Baseline | Pro-ocular + Placebo at 2 Years
Number analyzed (Participants) | 33 | 21
score on a scale | 3.67 (2.354) | 0.46 (0.886)
Statistical Analysis 1: Comparison: Pro-ocular + Placebo Baseline vs Pro-ocular + Placebo at 2 Years; Test type: Other; p < 0.00001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 2 years
Description: The entire study period of 2 years include a masked phase of 10 weeks, after which all participants received active drug for the remaining 2 years.
Groups:
- Pro-ocular™ for 2 Years: Pro-ocular™ 1% topical gel applied to forehead twice daily
- Pro-ocular™ for 10-week Masked Period Only: Pro-ocular™ 1% topical gel applied to forehead twice daily for 10-week masked period only
- Placebo+Active for 2 Years Total: Placebo topical gel applied to forehead twice daily. Placebo gel for the first 10 weeks of masked period, followed by active gel for the remaining 2 year period
- Placebo for 10-week Masked Period Ony: Placebo topical gel applied to forehead twice daily. Placebo gel for the first 10 weeks of masked period only
Arm/Group | Pro-ocular™ for 2 Years | Pro-ocular™ for 10-week Masked Period Only | Placebo+Active for 2 Years Total | Placebo for 10-week Masked Period Ony
All-Cause Mortality (participants affected / at risk) | 1/22 | 0/22 | 1/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 8/22 | 0/22 | 7/11 | 2/11
Other Adverse Events (participants affected / at risk) | 21/22 | 17/22 | 11/11 | 8/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pro-ocular™ for 2 Years (N=22) | Pro-ocular™ for 10-week Masked Period Only (N=22) | Placebo+Active for 2 Years Total (N=11) | Placebo for 10-week Masked Period Ony (N=11)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute lymphocytic leukaemia recurrent (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Endocrine neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular operation (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip surgery (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnea (Cardiac disorders) | 1 (1) | NA | 0 (0) | 0 (0)
Rib fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiopulmonary failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Corneal perforation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Corneal thinning (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal epithelium defect (Eye disorders) | 0 (0) | NA | 1 (3) | 0 (0)
Mycardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Cerebrovascular accident (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neurosensory hypoacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ophthalmic herpes simplex (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Corneal infiltrates (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parathyroidectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pro-ocular™ for 2 Years (N=22) | Pro-ocular™ for 10-week Masked Period Only (N=22) | Placebo+Active for 2 Years Total (N=11) | Placebo for 10-week Masked Period Ony (N=11)
Headache (Nervous system disorders) | 6 (6) | 6 (6) | 1 (1) | 1 (1) — Headaches were light and brief, lasting 10 min to 2 hours, occurring within the first 2 weeks of the study only.
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 6 (11) | 6 (11) | 0 (0) | 0 (0) — Rhinorrhea or runny nose in almost all cases were brief, and occurred within the first 2 weeks of the study only.
Conjunctival haemorrhage (Eye disorders) | 2 (3) | 1 (2) | 0 (0) | 0 (0)
Corneal abrasion (Eye disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 2 (2) | 2 (2) | 2 (2)
Eye pruritus (Eye disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Discomfort (General disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (2) | 1 (2) | 1 (2) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has prior review rights before publications or presentations.

DOCUMENTS (2):
  • Study Protocol (2020-03-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT03990051/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/51/NCT03990051/SAP_001.pdf